CLINICAL TRIAL: NCT00467545
Title: An Extension to A Randomized, Open-label, Controlled, Multicenter, Exploratory Trial to Characterize the Results of Daily Oral Administration of Telbivudine (LDT600) 600 mg or Entecavir (ETV) 0.5 mg Given Over 12 Weeks on the Kinetics of Hepatitis B Virus (HBV) DNA in Adults With HBeAg-positive, Compensated Chronic Hepatitis B (CHB) (An Open-label Multicenter, follow-on Trial of the Safety of Oral Administration of Telbivudine (LDT600) 600 mg Over 21 Months in Adults With HBeAg-positive Ompensated Chronic Hepatitis B (CHB))
Brief Title: An Extension to Viral Kinetics Study of Telbivudine and Entecavir in Adults With Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AKR02
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2012-05

CONDITIONS: Chronic Hepatitis B
Keywords: HBeAg-positive; chronic hepatitis B; telbivudine
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

INTERVENTIONS:
Drug: telbivudine

SUMMARY:
This study is to evaluate the safety of telbivudine for up to 21 months of open-label treatment in patients with chronic hepatitis B who have completed the CLDT600A2407 trial. Patients treated with telbivudine during core phase will continue telbivudine and patients treated with entecavir during core phase will be switched to telbivudine if the patient is willing to enroll this study.

ELIGIBILITY:
Inclusion Criteria:

* The patient has completed the previous CLDT600A2407 study and is able to immediately enter this extension study with no study drug discontinuation
* Patient is willing and able to comply with the study drug regimen and all other study requirements
* The patient is willing and able to provide written informed consent to participate in the extension study.

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient is co-infected with HCV, HDV, or HIV.
* History of malignancy of any organ system, treated or untreated, within the past 5 years with the exception of localized basal cell carcinoma of the skin.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety of telbivudine (LDT600) up to 21 additional months of open-label treatment in patients with chronic hepatitis B who have completed study CLDT600A2407 assessed by Adverse Events, data of vital signs and other tests

SECONDARY OUTCOMES:
Safety of patients switched from entecavir to telbivudine compared with patients continuing telbivudine assessed by Adverse Events, data of vital signs and other tests

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (6):
- South Korea (6):
  - Novartis Investigative Site (705-035), Daegu
  - Novartis Investigative Site , (420-717), Gyeonggi-do
  - Novartis Investigative Site , (405-760), Incheon
  - Novartis Investigative Site , (136-705), Seoul
  - Novartis Investigative Site , (150-590), Seoul
  - Novartis Investigative Site, Seoul